CLINICAL TRIAL: NCT06214234
Title: Timing of Upper Endoscopy in Cirrhotic Patients With Upper Gastrointestinal Bleeding: Urgent vs. Elective Endoscopy
Brief Title: Upper Endoscopy in Cirrhotic Patients With Upper Gastrointestinal Bleeding
Acronym: Varices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shadn Ahmed Keilany, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Shadn Protocol
Record Dates: First submitted 2024-01-08; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Varices
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Intervention Model Description: Two groups of patients present with variceal bleeding
Who Masked: Investigator
Masking Description: Patient will be enrolled in one each group without masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early band ligation (Other): Patients with liver cirrhosis present with variceal bleeding underwent band ligation within 12 hours of presentation
  Interventions: Procedure: Band ligation
- Delayed band ligation (Other): Patients with liver cirrhosis present with variceal bleeding underwent band ligation within more than 12 hours of presentation
  Interventions: Procedure: Band ligation

INTERVENTIONS:
Procedure: Band ligation — Band ligation in variceal bleeding

SUMMARY:
Liver cirrhosis is a common diffuse and persistent liver disease often accompanied by portal hypertension, liver failure, upper gastrointestinal bleeding (UGIB), and other complications. The incidence rate of liver cirrhosis with UGIB is as high as 30-40%, which is related to the rupture bleeding of gastroesophageal varices (GOV), hepatogenic ulcer, portal hypertensive gastropathy, hepatic gastrointestinal failure, etc

DETAILED DESCRIPTION:
In the case of UGIB in patients with liver cirrhosis, acute peripheral circulatory failure may suddenly occur, resulting in decreased blood perfusion in liver tissues, often accompanied by clinical manifestations such as blood volume decline, melena, and haematemesis. This disease progresses rapidly, with a mortality rate of above 10% if not treated promptly

Timing of endoscopy in the management of acute upper gastrointestinal bleeding (AUGIB) has been a subject of perennial debate. Despite remarkable advancements in endoscopic treatments and substantial efforts in reducing mortality, the overall in-hospital mortality rate associated with UGIB is still estimated to be 10%.

Several studies have investigated the clinical impact of urgent (within 6 h of presentation) or early (within 12 h) endoscopy on mortality in patients with UGIB. Some studies showed no significant difference in mortality rate between urgent and elective endoscopy groups among high-risk patients with acute UGIB

In contrast, others found that urgent endoscopy was associated with a lower mortality rate in high-risk patients with acute non-variceal UGIB. Most of the previous studies included highly selected patients with non-variceal UGIB or those at a high risk. However, given that the definitive diagnosis is made after endoscopic examination, these studies may not reflect real-world clinical practice. Furthermore, it is often challenging to predict the cause of bleeding and to identify patients at high risk who require intensive care based on their symptoms and the information obtained in the emergency room

ELIGIBILITY:
Inclusion Criteria:

Any patient who is above age of 18 years old and with liver cirrhosis and present with UGIB will be eligible for the study

Exclusion Criteria:

* Patients with age less than 18 years old
* Non-cirrhotic patients
* Patients with hemodynamic instability
* Patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
in-hospital bleeding | One year
  Frequency of mortality in patients with variceal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Shaden Kelany, MSc, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim J, Gong EJ, Seo M, Park JK, Lee SJ, Han KH, Kim YD, Jeong WJ, Cheon GJ, Seo HI. Timing of endoscopy in patients with upper gastrointestinal bleeding. Sci Rep. 2022 Apr 27;12(1):6833. doi: 10.1038/s41598-022-10897-3. PMID 35477727